CLINICAL TRIAL: NCT00712166
Title: A Double-Blind, Multicenter, Multinational, Randomized, Placebo-Controlled Trial Evaluating Aztreonam Lysine For Inhalation in Patients With Cystic Fibrosis, Mild Lung Disease, and P. Aeruginosa (AIR-CF4)
Brief Title: Safety and Efficacy Study of Aztreonam for Inhalation Solution (AZLI) in Patients With Cystic Fibrosis, Mild Lung Disease, and P. Aeruginosa
Acronym: AIR-CF4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Mark Bresnik, MD, Director, Clinical Research, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-205-0117
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-11

CONDITIONS: Cystic Fibrosis; Lung Infection; Pseudomonas Aeruginosa
Keywords: cystic fibrosis; pseudomonas aeruginosa; lung infection; CFQ-R; inhaled antibiotic; aztreonam lysine
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo three times daily (TID) (Placebo Comparator)
  Interventions: Drug: Placebo three times daily (TID)
- AZLI 75 mg three times daily (TID) (Experimental)
  Interventions: Drug: AZLI 75 mg three times daily (TID)

INTERVENTIONS:
Drug: AZLI 75 mg three times daily (TID)
  Arms: AZLI 75 mg three times daily (TID)
Drug: Placebo three times daily (TID)
  Arms: Placebo three times daily (TID)

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of a 28-day course of aztreonam for inhalation solution (AZLI) in patients with cystic fibrosis (CF), mild lung disease (forced expiratory volume in 1 second [FEV1] >75% predicted, and Pseudomonas aeruginosa (PA) infection.

DETAILED DESCRIPTION:
CF patients often have lung infections that occur repeatedly or worsen over time. The lung infections are often caused by a bacteria called Pseudomonas aeruginosa (PA). Treatment with antibiotics can stop or slow down the growth of the bacteria. The antibiotics may be given by mouth, intravenously (IV), or by inhalation as a mist. The purpose of this study was to evaluate the safety and efficacy of AZLI, an investigational formulation of the antibiotic aztreonam and administered three times a day using the PARI eFlow® electronic nebulizer, in CF patients with PA and mild lung disease.

In this study, participant eligibility was assessed at a screening visit that occurred up to 14 days prior to the baseline visit (Day 0). Those participants who met eligibility criteria at Day 0 were randomized and began a 28-day course of blinded study treatment (AZLI or placebo TID). Participants returned for clinic visits at Day 14, an end of treatment visit at Day 28, and a follow up visit 14 days after the last dose of the trial drug (Day 42).

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 6 years of age
* Documentation of CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

  * Sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test
  * Two well characterized mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
  * Abnormal nasal potential difference
* PA present in expectorated sputum or throat swab culture at Visit 1 OR documented PA in 2 expectorated sputum or throat swab cultures within the 12 months prior to Visit 1 (one of the previous PA positive cultures must have been no more than 3 months prior to Visit 1)
* FEV1 > 75% predicted at Visit 1
* Participants must have exhibited two or more of the following chronic and/or intermittent CF symptoms, for a minimum of 28 days prior to randomization and with no worsening of symptoms within 7 days prior to randomization:

  * Chest congestion
  * Daily cough
  * Productive cough
  * Wheezing
  * Trouble breathing
  * Nocturnal wakening due to coughing
* Participants (and parent/guardian as required) had to be able to provide written informed consent/assent prior to any study related procedures
* Females of childbearing potential had to have a negative urine pregnancy test at Visit 1
* Ability to perform reproducible pulmonary function tests
* In the opinion of the Investigator, the participant did not require immediate antipseudomonal antibiotic intervention to treat an impending exacerbation, and the participant's condition was stable enough to enroll in the study

Exclusion Criteria:

* Administration of any investigational drug or device within 28 days prior to Visit 1 or within 6 half-lives of the investigational drug (whichever was longer)
* Administration of any IV, oral, or inhaled antipseudomonal antibiotic within 28 days prior to Visit 1
* Known local or systemic hypersensitivity to monobactam antibiotics
* Inability to tolerate short-acting bronchodilator (BD) use at least TID
* Changes in or initiation of chronic azithromycin treatment within 28 days prior to Visit 1
* Changes in or initiation of chronic hypertonic saline treatment within 28 days prior to Visit 1
* Changes in or initiation of dornase alfa within 28 days prior to Visit 1
* Changes in antimicrobial, BD, or corticosteroid medications within 7 days prior to Visit 1
* Changes in physiotherapy technique or schedule within 7 days prior to Visit 1
* History of lung transplantation
* History of participation (enrollment) in any prior clinical studies with AZLI
* A chest radiograph at Visit 1 (or within the previous 180 days of Visit 1), with abnormalities indicating a significant acute finding (e.g., lobar infiltrate and atelectasis, pneumothorax, or pleural effusion); a chest radiograph obtained and interpreted between Visits 1 and 2 was also acceptable for determining eligibility
* Positive urine pregnancy test at Visit 1; all women of childbearing potential were to be tested
* Females of childbearing potential who were lactating or were not (in the opinion of the investigator) practicing an acceptable method of birth control; female participants who utilized hormonal contraceptives as their birth control method must have used the same method for at least 3 months before study dosing
* Participant was being assessed at Visit 1 by the investigator for an acute change in respiratory symptoms
* Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would have interfered with participant treatment, assessment, or compliance with the protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Wainwright, MD, Principal Investigator — Royal Children's Hospital, Brisbane, QLD, Australia; Ron Gibson, MD, Principal Investigator — Children's Hospital & Regional Medical Center, Seattle WA, USA
Locations (40):
- United States (34):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Division of Pulmonary and Critical Care Medicine, Little Rock, Arkansas
  - Kaiser Permanente, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - The Children's Hospital, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Indiana University, Outpatient Clinical Research Facility, Indianapolis, Indiana
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital, Boston, Boston, Massachusetts
  - Tufts Medical Center, Pediatric Pulmonary Clinic, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - The Children's Hospital of Michigan, Detroit Medical Center, Detroit, Michigan
  - The Minnesota CF Center, University of Minnesota Medical Center, Minneapolis, Minnesota
  - Children's Lung Specialists, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - The Lung & Cystic Fibrosis Center, University of Buffalo Pediatric Associates, Inc., Women & Children's Hospital of Buffalo, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital/Toledo Hospital, Cystic Fibrosis Research Center, Toledo, Ohio
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Pulmonary Associates, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- Australia (5):
  - Department of Respiratory Medicine, The Children's Hospital at Westmead, Westmead, New South Wales
  - Department of Respiratory Medicine, Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Adult Cystic Fibrosis Centre, Chermside, Queensland
  - Respiratory Medicine, Royal Children's Hospital, Herston, Queensland
  - Child and Adolescent Health Services, Princess Margaret Hospital, Perth, Western Australia
- Centre de Recherche du CHUM, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Wainwright CE, Quittner AL, Geller DE, Nakamura C, Wooldridge JL, Gibson RL, Lewis S, Montgomery AB. Aztreonam for inhalation solution (AZLI) in patients with cystic fibrosis, mild lung impairment, and P. aeruginosa. J Cyst Fibros. 2011 Jul;10(4):234-42. doi: 10.1016/j.jcf.2011.02.007. Epub 2011 Mar 26. PMID 21441078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 39 sites in total: 34 in the United States, 1 in Canada, and 4 in Australia. Date of first screening was 16 June 2008, and date of last participant observation was 19 June 2009.
Pre-assignment Details: Planned trial size was approximately 140 participants randomized in 1:1 ratio to aztreonam for inhalation solution (AZLI) three times daily (TID) or placebo TID. 160 participants were randomized, 157 received blinded study drug (76 AZLI; 81 placebo). One participant who was randomized and treated with study drug discontinued the study.
Groups:
- Placebo Three Times Daily (TID): Placebo (5 mg/mL lactose when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.5, and osmolality 200 to 400 mOsmol/kg). Placebo was self-administered TID by inhalation using the investigational nebulizer.
- AZLI 75 mg Three Times Daily (TID): AZLI (75 mg/mL aztreonam lysine when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.0, and osmolality 300 to 550 mOsmol/kg). AZLI was self-administered by inhalation TID using the investigational nebulizer.
Period: Overall Study
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Started | 81 | 76
Completed | 81 | 75
Not Completed | 0 | 1
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID) | Total
Number analyzed (Participants) | 81 | 76 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 42 | 89
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 18.9 (9.11) | 19.5 (9.07) | 19.2 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 30 | 67
  Male | 44 | 46 | 90
Region of Enrollment [Number; unit: participants]
  United States | 73 | 72 | 145
  Canada | 2 | 0 | 2
  Australia | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS) Score at Day 28
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for children and adults with CF. The CFQ-R contains both general and CF-specific scales. The CFQ-R was administered at Days 0, 14, 28, and 42. The endpoint was change in respiratory symptoms (e.g., coughing, congestion, wheezing) from Day 0 (baseline), assessed with the CFQ-R RSS (score range: 0-100; higher scores indicating fewer symptoms, higher health-related quality of life, or better functioning). Baseline CFQ-R RSS and age group (<18 vs. >=18 years) were included as covariates in the analysis.
Time Frame: Day 0 to Day 28
Population: Analysis on intent-to-treat (ITT) population (received at least part of 1 dose of AZLI/placebo). Missing baseline data not imputed. Missing post-baseline data imputed with worst-case value for participants who withdrew due to an adverse event (AE)/study drug intolerance. Imputation for other missing data was last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Units on a scale | 1.41 (1.64) | 3.22 (1.71)
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in CFQ-R RSS score at Day 28. At the 5% significance level (i.e., α = 0.05) using a two-sided significance test, a sample size of 70 participants per treatment group provided at least 90% power to detect a 10 point difference between groups in the mean change from baseline at Day 28 in the CFQ-R RSS score, assuming a common standard deviation (SD) of 17.5; Test type: Superiority or Other; p = 0.433, ANCOVA — The primary endpoint analysis was based on a two-sided test with an 0.05 a priori threshold for statistical significance. A gate-keeper approach was established a priori to control the type 1 error rate, however, the primary endpoint was not met; ANCOVA included: treatment, baseline CFQ-R RSS, age group (<18, >=18 years). Denominator degrees of freedom computed with Satterthwaite approximation; Mean Difference (Final Values) = 1.80, 95% CI 2-sided [-2.83 to 6.44]

2. Secondary Outcome: Change From Baseline in CFQ-R RSS Score at Day 14
Description: as for outcome 1
Time Frame: Day 0 to Day 14
Population: Analysis based on ITT population (all participants receiving at least part of one dose of AZLI or placebo). Missing baseline data were not imputed. Missing post-baseline data were imputed using worst-case value for participants who withdrew due to an AE or study drug intolerance. For all other missing data, LOCF imputation method was used.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Units on a scale | 0.28 (1.56) | 3.65 (1.63)
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in the CFQ-R RSS score at Day 14; Test type: Superiority or Other; p = 0.133, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA included terms: treatment, baseline CFQ-R RSS, age group (<18, >=18 years). Treatment differences were calculated as AZLI-placebo; Mean Difference (Final Values) = 3.37, 95% CI 2-sided [-1.04 to 7.78]

3. Secondary Outcome: Change From Baseline in CFQ-R RSS Score at Day 42
Description: as for outcome 1
Time Frame: Day 0 to Day 42
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Units on a scale | 2.91 (1.65) | 3.02 (1.72)
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in the CFQ-R RSS score at Day 42; Test type: Superiority or Other; p = 0.965, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included terms for treatment, baseline CFQ-R RSS and age group (<18 years, >=18 years). Treatment differences calculated as AZLI-placebo; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-4.56 to 4.76]

4. Secondary Outcome: Change From Baseline in CFQ-R Physical Functioning Domain Score
Description: The CFQ-R contains both general and CF-specific scales. The CFQ-R was administered at Days 0 (baseline), 14, 28, and 42 (the last study visit). The endpoint was change from baseline in the physical functioning domain (e.g., ability to walk and engage in physical activities) of the CFQ-R at Day 28 (range of scores: 0-100; higher scores indicating fewer symptoms, higher health-related quality of life, or better functioning). Baseline CFQ-R physical functioning domain score and age group (<18 vs. >=18 years) were included as covariates in the analysis.
Time Frame: Day 0 to Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Units on a scale | -0.69 (1.53) | 1.79 (1.57)
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in the CFQ-R physical functioning domain score at Day 28; Test type: Superiority or Other; p = 0.256, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA included: treatment, baseline CFQ-R Physical Function Domain score and age (<18, >=18 years). Treatment differences calculated as AZLI-placebo; Mean Difference (Final Values) = 2.47, 95% CI [-1.81 to 6.76]

5. Secondary Outcome: Number of Participants Using Additional (Nonprotocol-specified) Antipseudomonal Antibiotics During Study
Description: The number of participants requiring additional antipseudomonal antibiotics (oral, intravenous [IV], or by inhalation), the time to use of these antibiotics, and the reasons for use was recorded. A binary variable was defined to indicate whether the participants needed any antipseudomonal antibiotics that were non-study drug via the oral, IV, or inhalation route between Day 0 (Baseline Visit) and Day 42 (Visit 5). Fisher's Exact Test was implemented on the intent-to-treat (ITT) and per protocol analysis sets to detect treatment effects on need for additional antipseudomonal antibiotics.
Time Frame: Day 0 to Day 42
Population: Analysis based on ITT population (all participants who received at least part of one dose of AZLI or placebo). No imputation methods were used for the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Participants | 21 | 19
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in number of participants using additional (nonprotocol-specified) antipseudomonal antibiotics during study; Test type: Superiority or Other; p > 0.999, Fisher Exact — No adjustments were made for multiple comparisons; A participant with multiple usage was counted only once

6. Secondary Outcome: Number of Participants Hospitalized During Study
Description: Hospitalization was defined as any hospital admission lasting for more than 1 calendar day that had been recorded as a serious adverse event (SAE) on the electronic case report form (eCRF). Binary variables were defined to indicate whether participants experienced any hospitalization. Number of hospitalizations was summarized by treatment group.
Time Frame: Day 0 to Day 42
Population: as for outcome 5
Measure: Number; unit: Study participants
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Study participants | 3 | 8
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in proportion of participants hospitalized; Test type: Superiority or Other; p = 0.122, Fisher Exact — No adjustments were made for multiple comparisons; A participant with multiple hospitalizations was counted only once

7. Other Pre Specified Outcome: Number of Participants Testing Positive for Other Respiratory Pathogens
Description: Sputum/throat swab samples were collected at all visits for quantitative and qualitative culture of Burkholderia species, Stenotrophomonas maltophilia, Achromobacter xylosidans, methicillin-resistant Staphylococcus aureus (MRSA), methicillin-sensitive S. aureus (MSSA), and Aspergillus species. One CFU on the culture from either a sputum or throat swab sample was considered presence of the particular organism.
Time Frame: Day 0 to Day 28
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Participants
  B. cepacia - Day 0 | 1 | 0
  B. cepacia - Day 28 | 1 | 1
  S. maltophilia - Day 0 | 7 | 8
  S. maltophilia - Day 28 | 9 | 8
  A. xylosoxidans - Day 0 | 0 | 1
  A. xylosoxidans - Day 28 | 2 | 1
  MRSA - Day 0 | 14 | 14
  MRSA - Day 28 | 13 | 13
  MSSA - Day 0 | 31 | 28
  MSSA - Day 28 | 31 | 25
  Aspergillus spp. - Day 0 | 6 | 10
  Aspergillus spp. - Day 28 | 6 | 11

8. Other Pre Specified Outcome: The Minimum Concentrations of Aztreonam That Inhibit 50% and 90% of All PA Isolates (MIC50 and MIC90, Respectively)
Description: Aztreonam susceptibility of PA isolates from expectorated sputum samples (collected at all visits) was assessed. The minimum inhibitory concentration (MIC) is the lowest concentration of antimicrobial agent that inhibits visible growth of a microorganism. The MIC50 and MIC90 for PA is the MIC required to inhibit the growth of 50% or 90% of PA isolates, respectively. Given that there might be multiple PA isolates for each participant, the MIC50 and MIC90 for PA was calculated using the MIC values for all PA isolates. The MIC50 and MIC90 were calculated by treatment group.
Time Frame: Day 0 to Day 28
Population: Analysis based on ITT population (all participants who received at least part of one dose of AZLI or placebo).
Measure: Number; unit: µg/mL
Groups:
- Placebo TID: Placebo (5 mg/mL lactose when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.5, and osmolality 200 to 400 mOsmol/kg). Placebo was self-administered TID by inhalation using the investigational nebulizer.
  Day 0: number of isolates = 104; Day 28: number of isolates = 108
- AZLI 75 mg TID: AZLI (75 mg/mL aztreonam lysine when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.0, and osmolality 300 to 550 mOsmol/kg). AZLI was self-administered by inhalation TID using the investigational nebulizer.
  Day 0: number of isolates = 104; Day 28: number of isolates = 76
Arm/Group | Placebo TID | AZLI 75 mg TID
Number analyzed (Participants) | 81 | 76
µg/mL
  Baseline MIC50 | 1 | 1
  Day 28 MIC50 | 1 | 4
  Baseline MIC90 | 16 | 8
  Day 28 MIC90 | 16 | 32

9. Secondary Outcome: Change From Baseline in Log10 Pseudomonas Aeruginosa (PA) Colony Forming Units (CFUs) in Sputum at Day 28
Description: Sputum samples were collected at all study visits for quantitative and qualitative culture for PA. Sputum PA density was quantified by logarithm transformation of the CFU value with base 10. Change from baseline in sputum PA density was calculated as the difference between the log10 CFU values at Day 28 (Visit 4) and the baseline value. Missing data was not imputed. Baseline log10 CFU and age group (<18 vs. >=18 years) were included as covariates in the analysis.
Time Frame: Day 0 to Day 28
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Log10 PA CFUs/gram of sputum
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 31 | 37
Log10 PA CFUs/gram of sputum | -0.14 (0.36) | -1.35 (0.36)
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in change from baseline in the log10 CFU at Day 28; Test type: Superiority or Other; p = 0.016, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included treatment, baseline log10 CFU, and age group (<18, >=18 years). Treatment differences were calculated as AZLI-placebo; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-2.20 to -0.23]

10. Secondary Outcome: Relative Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted
Description: Spirometry was performed according to American Thoracic Society (ATS) guidelines at each visit. Treatment effect on the relative change from baseline in FEV1 percent predicted at Day 28 (Visit 4) was tested by the ANCOVA model using the ITT analysis set. Baseline FEV1 percent predicted and age group (<18 vs. >=18 years) were included as covariates in the analysis.
Time Frame: Day 0 to Day 28
Population: Analysis based on ITT population (all participants who received at least part of one dose of AZLI or placebo). Missing baseline data were not imputed. Missing post-baseline data were imputed using worst-case value for participants who withdrew due to an AE or study drug intolerance. For all other missing data, LOCF method was used.
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Number analyzed (Participants) | 81 | 76
Percent change from baseline | -2.45 (0.82) | 0.29 (0.85)
Statistical Analysis 1: Comparison: Placebo Three Times Daily (TID) vs AZLI 75 mg Three Times Daily (TID); Null hypothesis was there was no difference between 75 mg AZLI TID and placebo treatment groups in % change from baseline in FEV1 % predicted at Day 28; Test type: Superiority or Other; p = 0.021, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model includes treatment, baseline FEV1 % predicted, and age group (<18, >=18 years). Treatment differences were calculated as AZLI-placebo; Mean Difference (Final Values) = 2.73, 95% CI 2-sided [0.42 to 5.04]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected continuously from the first dose (Day 0) until 14 days after last AZLI/placebo dose (typically Day 42). Participants who discontinued were evaluated for at least 14 days after last dose of study drug.
Description: An AE was any physical/clinical worsening in symptoms/disease (including clinically significant change in lab values) experienced by participant at any time during study, whether or not event was considered related to study participation or study procedures. Participants were only counted once within a System Organ Class (SOC) and preferred term.
Arm/Group | Placebo Three Times Daily (TID) | AZLI 75 mg Three Times Daily (TID)
Serious Adverse Events (participants affected / at risk) | 3/81 | 9/76
Other Adverse Events (participants affected / at risk) | 62/81 | 58/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Three Times Daily (TID) (N=81) | AZLI 75 mg Three Times Daily (TID) (N=76)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pseudomonas bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Three Times Daily (TID) (N=81) | AZLI 75 mg Three Times Daily (TID) (N=76)
Abdominal pain (Gastrointestinal disorders) | 9 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 32
Decreased appetite (Metabolism and nutrition disorders) | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Dizziness (Nervous system disorders) | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Fatigue (General disorders) | 10 | 6
Headache (Nervous system disorders) | 10 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Nausea (Gastrointestinal disorders) | 6 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 | 18
Pulmonary function test decreased (Investigations) | 8 | 6
Pyrexia (General disorders) | 7 | 5
Rales (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.